CLINICAL TRIAL: NCT03648541
Title: An Open Label, Long Term Safety Trial of BI 655130 (SPESOLIMAB) Treatment in Patients With Moderate to Severely Active Ulcerative Colitis Who Have Completed Previous BI 655130 Trials
Brief Title: BI 655130 Long-term Treatment in Patients With moderate-to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0017; 2018-000334-35 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab IV infusion (Experimental): Spesolimab IV infusion
  Interventions: Drug: Spesolimab
- Spesolimab SC solution for injection (Experimental): Spesolimab SC solution for injection
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Solution

SUMMARY:
To evaluate the long-term safety of BI 655130 (SPESOLIMAB) in patients with moderate to severely active ulcerative colitis, who have completed treatment in previous trials

To evaluate the long-term efficacy of BI 655130 (SPESOLIMAB) in patients with moderate to severely active ulcerative colitis, who have completed treatment in previous trials

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged ≥18 years
* Signed and dated written informed consent for 1368.17, in accordance with GCP and local legislation prior to admission into the trial
* Women of childbearing potential (WOCBP) must be ready to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. Note: A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tuba ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Have completed treatment and the EOT visit in the previous trial and are willing and able to continue treatment in 1368.17.

Exclusion Criteria:

* Have experienced study treatment-limiting adverse events during induction treatment with study drug
* Have developed any of the exclusion criteria from the original induction study with the following exceptions:

  * Cases of disease limited to the rectum extending <15 cm past the anal verge are allowed to be included in study 1368.17
  * Cases of latent TB. Patients with newly emerging latent TB during preceding study are allowed to be included in study 1368.17, provided they receive appropriate treatment according to local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (8):
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
- Austria (2):
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - AKH - Medical University of Vienna, Vienna
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Victoria Hospital (LHSC), London, Ontario, Canada
- Germany (6):
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Asklepios Kliniken Westklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Istituto Clinico Humanitas, Rozzano (MI)
- Japan (6):
  - Sapporo Tokushukai Hospital, Hokkaido, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Hokkaido, Sapporo
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - Ofuna Chuo Hospital, Kanagawa, Kamakura
  - Tokyo Medical and Dental University Hospital, Tokyo, Bunkyo-ku
  - Tokyo Yamate Medical Center, Tokyo, Shinjuku
- National Medical Institute MSWiA, Warsaw, Poland
- Russia (3):
  - FSB Instit. HC Irkutsk Scient.Cent. Sibirian Branch of Russ. Acad. Scien., Irkutsk
  - Federal State Budgetary Institution " State Scientific Center of Coloproctology" MOH Russia, Moscow
  - Military Medical Academy n.a. C. M. Kirov, St. Petersburg, Saint Petersburg
- South Korea (2):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
- Spain (2):
  - Hospital Virgen del Rocío, Seville
  - Hospital Politècnic La Fe, Valencia
- United Kingdom (3):
  - Doncaster Royal Infirmary, Doncaster
  - Guy's Hospital, London
  - Whiston Hospital, Prescot

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label 7-year long-term extension trial in patients with moderate-to-severe ulcerative colitis who completed treatment in previous spesolimab trials 1368-0005 (NCT03482635) Part 1 and 1368-0004 (NCT03100864).
Pre-assignment Details: Only subjects that met the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all subjects as required.
Groups:
- 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks: Participants who completed treatment in the parent trial, but did not have a clinical response at Week 12 (end of trial (EOT)), entered a 12-week spesolimab re-induction period, receiving multiple active doses of 1200 milligrams (mg) solution for infusion of spesolimab as intravenous (i.v.) infusion every 4 weeks (q4w) for 12 weeks (re-induction). If participants reached a clinical response at Week 12 of the re-induction treatment, they switched to the maintenance treatment receiving 300 mg solution of injection of spesolimab as subcutaneous (s.c.) injection q4w for up to 336 weeks. Participants who did not achieve a clinical response after 12 weeks of re-induction treatment were discontinued from treatment.
- 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks: 300 mg solution for injection of spesolimab was administered as subcutaneous (s.c.) injection q4w for 336 weeks as maintenance treatment.
  This arm included participants who entered the maintenance treatment directly from the parent trial and participants who switched from the re-induction treatment.
  Participants who completed treatment in the parent trial and had a clinical response at week 12 (EOT) directly received maintenance treatment. Participants, who started re-induction treatment, could switch to maintenance treatment if they reached a clinical response at Week 12 of the re-induction period.
  Participants who experienced a disease flare during maintenance treatment were administered a single intravenous dose of spesolimab 1200 mg followed by an intensified subcutaneous maintenance dosing schedule with 600 mg q6w.
Period: Started From Parent Trial
Arm/Group | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
Started (Number of participants from parent trials who were enrolled into 1368-0017.) | 57 (Number of participants from parent trial who received re-induction treatment.) | 22 (Number of participants from parent trial who directly received maintenance treatment.)
Completed (Completed reflects the number of participants who either started re-induction period or maintenance period or both.) | 57 | 22
Not Completed | 0 | 0
Period: Re-induction Period Only
Arm/Group | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
Started (Started re-induction treatment.) | 57 | 0
Switched to Maintenance Treatment | 12 | 0
Completed (Completed re-induction treatment.) | 49 | 0
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Efficacy | 7 | 0
Period: Maintenance Period Only
Arm/Group | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
Started (Started maintenance treatment) | 0 | 34
Participants From Parent Trial | 0 | 22
Participants From Re-induction Treatment | 0 | 12
Completed (Completed maintenance treatment) | 0 | 0
Not Completed | 0 | 34
Not completed — Missing | 0 | 1
Not completed — Other not listed below | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 18
Not completed — Adverse Event | 0 | 4
Not completed — Stopped maintenance treatment due to study stop | 0 | 3

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose on maintenance or re-induction treatment in the extension trial.
  Baseline characteristics are reported for maintenance treatment and re-induction treatment combined, as these arms are not mutually exclusive and patients could switch from re-induction treatment to maintenance treatment.
Groups:
- Spesolimab - All Patients: Patients with moderate-to-severe ulcerative colitis who completed treatment in previous spesolimab induction trials. Patients were treated according to their previous trial outcome. Those who completed treatment in the previous trials showing a clinical response (CR) directly received maintenance treatment, consisting of 300 mg solution for injection of spesolimab administered as subcutaneous (s.c.) injection q4w for 336 weeks. Patients who did not achieve a clinical response in the previous trials received multiple active doses of 1200 milligrams (mg) solution for infusion of spesolimab as intravenous (i.v.) infusion every 4 weeks (q4w) for 12 weeks, as re-induction treatment. If participants reached a clinical response at Week 12 of the re-induction treatment, they switched to the maintenance treatment receiving 300 mg solution of injection of spesolimab as subcutaneous (s.c.) injection q4w for up to 336 weeks.
Arm/Group | Spesolimab - All Patients
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Exposure Adjusted Rate of Participants Reporting a Treatment Emergent Adverse Event (TEAE)
Description: Exposure adjusted rate of participants reporting a treatment emergent adverse event (TEAE).
  The exposure adjusted incidence rate (per 100 subject years) of a selected treatment emergent adverse event is defined as the number of subjects experiencing the adverse event per treatment group during time at risk divided by the total time of subjects at risk in that treatment group to contribute the event to the analysis multiplied by 100 (per 100 subject years).
  Only participants receiving maintenance treatment were analysed for this endpoint.
Time Frame: From first maintenance treatment until last maintenance treatment, plus residual effect period (REP) of 112 days, up to 1550 days.
Population: SAF-MT: All participants who received at least one dose of maintenance treatment in this extension trial. Only participants receiving maintenance treatment were analysed for this endpoint.
Measure: Number; unit: Events per 100 patient-years
Arm/Group | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
Number analyzed (Participants) | 34
Events per 100 patient-years | 260.6

2. Secondary Outcome: Proportion of Patients With Clinical Remission at Week 336 of Maintenance Treatment
Description: Proportion of patients with clinical remission at Week 336 of maintenance treatment. Clinical remission was defined as rectal bleeding score (RBS) = 0, modified endoscopic subscore [mESS] ≤1, stool frequency score (SFS) = 0 or 1 and drop ≥1 from baseline, and modified mayo clinical score ((MCS) ≤2).
Time Frame: Up to 336 weeks
Population: Since this trial was prematurely ended and no patient achieved the Week 336 visit, no data satisfied the reporting criteria, and the endpoint could not be analysed.
Arm/Group | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Re-induction period: From first re-induction treatment until last re-induction treatment plus residual effect period (REP) of 112 days, up to 184 days for patients who did not participate in the maintenance treatment and from first re-induction treatment until first maintenance treatment minus 1 minute, up to 78 days for patients who continued with maintenance treatment. Maintenance period: From first maintenance treatment until last, plus REP of 112 days, up to 1550 days.
Description: (SAF-RT): All participants who received at least on dose of re-induction treatment in this extension trial; (SAF-MT): All participants who received at least on dose of maintenance treatment in this extension trial. Arms are not mutually exclusive.
Arm/Group | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks
All-Cause Mortality (participants affected / at risk) | 0/57 | 1/34
Serious Adverse Events (participants affected / at risk) | 3/57 | 6/34
Other Adverse Events (participants affected / at risk) | 14/57 | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks (N=57) | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks (N=34)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1200 mg Spesolimab i.v. Re-induction Treatment [q4w] for 12 Weeks (N=57) | 300 mg Spesolimab s.c. Maintenance Treatment [q4w] for 336 Weeks (N=34)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 9
Haemorrhoids (Gastrointestinal disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 5
Nasopharyngitis (Infections and infestations) | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 0 | 5
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anorectal discomfort (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3
COVID-19 (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Depression (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This trial was prematurely ended due to the decision to discontinue the clinical development of spesolimab in inflammatory bowel disease. This decision was based on a lower-than-expected efficacy in previous clinical trials conducted in ulcerative colitis and fistulising Crohn's disease. The decision was not related to any safety findings. The trial was completed as described in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT03648541/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03648541/SAP_001.pdf